CLINICAL TRIAL: NCT00000286
Title: Effects of Nefazodone on Treatment of Female Cocaine Abusers
Brief Title: Effects of Nefazodone on Treatment of Female Cocaine Abusers - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-3; P50-09259-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — nefazodone

INTERVENTIONS:
Drug: Nefazodone

SUMMARY:
The purpose of this study is to determine the effects of nefazedone on cocaine self-administration in depressed and non-depressed female cocaine users.

DETAILED DESCRIPTION:
This study evaluated the effect of nefazodone on reducing cocaine use and craving in both depressed and nondepressed women and if there was a greater effect in depressed women.

ELIGIBILITY:
Inclusion Criteria:

Females, ages 18-55, minimum use of 8 days of the last 30, minimum of 8th grade education, current diagnosis of cocaine abuse/dependence

Exclusion Criteria:

Unstable medical illness, dx of MR, OBS, bipolar

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-12; Study Completion 2001-12

PRIMARY OUTCOMES:
Craving
Drug use
Depression
Life functioning
HIV risk behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States